CLINICAL TRIAL: NCT04218474
Title: Evaluation Of Cross Mental Nerve Transfer In Restoration Of Lower Chin &Lip Sensation Post Inferior Alveolar Nerve Injury and Ablative Mandibular Resectons
Brief Title: Evaluation Of Cross Mental Nerve Transfer In Restoration Of Chin &Lip Sensation Post Inferior Alveolar Nerve Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmed Mohamed Basem (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohamed Basem, DR Ahmed Basem (Principle Investigator), Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2569369
Record Dates: First submitted 2019-11-27; First posted 2020-01-06 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Injury of Mental Nerve of One Side

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient lost sensation ant half of lower lip (Other): patient with injured inferior alveolar nerve at one side
  Interventions: Procedure: Evaluation Of Cross Mental Nerve Transfer In Restoration Of Chin &Lip Sensation Post Inferior Alveolar Nerve Injury

INTERVENTIONS:
Procedure: Evaluation Of Cross Mental Nerve Transfer In Restoration Of Chin &Lip Sensation Post Inferior Alveolar Nerve Injury — -sural nerve harvest ,and use it as conduit between injured mental nerve and the normal one

SUMMARY:
Evaluation Of Cross Mental Nerve Transfer In Restoration Of Chin &Lip Sensation Post Inferior Alveolar Nerve Injury

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemimandiblectomy
* Patients with Injured Inferior Alveolar Nerve which not showing any healing after 9 months
* Age group : from 15 to 60 years old
* No sex predilection
* Patients with no contraindications to surgical intervention

Exclusion Criteria:

* • Patients with systemic condition counteracting with the surgical procedure.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation Of Cross Mental Nerve Transfer In Restoration Of Chin &Lip Sensation Post Inferior Alveolar Nerve Injury | 1 year
  The primary outcome is restoration of sensation of lower lip and chin sensation determined by Two discrimination point test at 6 months . Aggregation will be done by percentage/ratio of successful cases number in the study. Calculation of the mean of all cases will be performed for analysis of the results.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kaban LB, Upton J. Cross mental nerve graft for restoration of lip sensation after inferior alveolar nerve damage: report of case. J Oral Maxillofac Surg. 1986 Aug;44(8):649-51. doi: 10.1016/s0278-2391(86)80078-7. No abstract available. PMID 3461143